CLINICAL TRIAL: NCT04226638
Title: Slipping Rib Syndrome: A Clinical Entity to Consider in Chest Pain
Status: Completed | Type: Observational
Sponsor: AMS Centro Medico del Ejercicio (Other)
Responsible Party: Principal Investigator, Carlos Leonardo Cano Herrera, Physiotherapy, AMS Centro Medico del Ejercicio
Other Study IDs: AMS CentroMédicoEjercicio
Record Dates: First submitted 2020-01-09; First posted 2020-01-13 (Actual); Last update posted 2020-01-13 (Actual); Status verified 2020-01

CONDITIONS: Slipping Rib Syndrome
Keywords: Slipping rib syndrome; dynamic ultrasound
MeSH Terms: conditions — Tietze's Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Dynamic ultrasound — Diagnosis was based on clinic suspicion and positive ultrasonography dynamic maneuvers by reproducing pain and slipping rib exam

SUMMARY:
Slipping rib syndrome consists on false or floating ribs hypermobility, whose can force the ribs to come in contact with each other. The authors reported a fourteen case series presenting a slipping rib syndrome.

DETAILED DESCRIPTION:
Slipping rib syndrome consists on false or floating ribs hypermobility, whose can force the ribs to come in contact with each other.

The authors reported a fourteen case series presenting a slipping rib syndrome. Mean age 35.00 ± 10.66 years old; 64.29% men.

The 10th rib level was the most predominant, affecting 64.29% of cases. Dynamic ultrasound was the gold standard diagnostic tool. Different conservative treatments were applied in most of cases.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting costal pain around 9th, 10th, or 11th rib.

Exclusion Criteria:

* Patients younger than 18 years old and older than 80 years old.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients affected with Slipping rib syndrome
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2017-02-02 (Actual); Primary Completion 2019-11-10 (Actual); Study Completion 2019-11-10 (Actual)

PRIMARY OUTCOMES:
Hypermobility level | 10 minutes
  Level of costal rib where there is hypermobility

SECONDARY OUTCOMES:
Sports | 1 minute
  If the subject participates in some kind of sport activity
Pain mechanism | 2 minutes
  Pain mechanism could be "repetitive movement", "trauma" or "pregnancy"
Diagnosis delay | 1 minute
  Time of delay in have a diagnosis (in years)

CONTACTS AND LOCATIONS:
Overall Officials: Ramón Balius, Principal Investigator — Consell Català de l'Esport. Generalitat de l'Esport. Barcelona. Spain.
Locations (1):
- DCR Trauma Group. Moreres Medical Center. Clínica Sagrada Família., Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Saltzman DA, Schmitz ML, Smith SD, Wagner CW, Jackson RJ, Harp S. The slipping rib syndrome in children. Paediatr Anaesth. 2001 Nov;11(6):740-3. doi: 10.1046/j.1460-9592.2001.00754.x. PMID 11696155
- [Background] Meuwly JY, Wicky S, Schnyder P, Lepori D. Slipping rib syndrome: a place for sonography in the diagnosis of a frequently overlooked cause of abdominal or low thoracic pain. J Ultrasound Med. 2002 Mar;21(3):339-43. doi: 10.7863/jum.2002.21.3.339. PMID 11883545
- [Background] Udermann BE, Cavanaugh DG, Gibson MH, Doberstein ST, Mayer JM, Murray SR. Slipping Rib Syndrome in a Collegiate Swimmer: A Case Report. J Athl Train. 2005 Jun;40(2):120-122. PMID 15970959
- [Background] Mooney DP, Shorter NA. Slipping rib syndrome in childhood. J Pediatr Surg. 1997 Jul;32(7):1081-2. doi: 10.1016/s0022-3468(97)90403-6. PMID 9247238
- [Background] Lum-Hee N, Abdulla AJ. Slipping rib syndrome: an overlooked cause of chest and abdominal pain. Int J Clin Pract. 1997 Jun;51(4):252-3. PMID 9287271
- [Background] Turcios NL. Slipping rib syndrome in an adolescent: an elusive diagnosis. Clin Pediatr (Phila). 2013 Sep;52(9):879-81. doi: 10.1177/0009922812469290. Epub 2012 Dec 12. No abstract available. PMID 23242850
- [Background] Bonasso PC, Petrus SN, Smith SD, Jackson RJ. Sternocostal slipping rib syndrome. Pediatr Surg Int. 2018 Mar;34(3):331-333. doi: 10.1007/s00383-017-4221-1. Epub 2017 Dec 6. PMID 29214341
- [Background] Van Tassel D, McMahon LE, Riemann M, Wong K, Barnes CE. Dynamic ultrasound in the evaluation of patients with suspected slipping rib syndrome. Skeletal Radiol. 2019 May;48(5):741-751. doi: 10.1007/s00256-018-3133-z. Epub 2019 Jan 5. PMID 30612161